CLINICAL TRIAL: NCT07096180
Title: Clinical Observational Studies: Breast Cancer Treatment by Traditional Chinese and Western Medicine
Brief Title: Clinical Observational Studies:Integrative TCM and Western Medicine for Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Principal Investigator, Hsien-Chang Wu, Director of the Department of Traditional Chinese Medicine, Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Other Study IDs: 12-XD-090
Record Dates: First submitted 2025-06-03; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: Traditional Chinese medicine; Adjunctive therapy; Side-Effect; Quality of Life
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional Western Medicine Treatment Group: Patients receive standard Western medical care, including chemotherapy, according to clinical guidelines. No Traditional Chinese Medicine (TCM) is involved. Clinical assessments and questionnaires are administered throughout the treatment course.
  Interventions: Drug: Chemotherapy drug
- Integrative Treatment Group (Western Medicine + TCM): Patients receive both standard Western medical care (e.g., chemotherapy) and Traditional Chinese Medicine (TCM) treatments. TCM is prescribed based on syndrome differentiation and focuses on supporting healthy qi and mitigating side effects. Clinical assessments and questionnaires are administered throughout the treatment course.
  Interventions: Other: Integrative Treatment (Chemotherapy + TCM)

INTERVENTIONS:
Drug: Chemotherapy drug — Participants in the standard care group receive conventional chemotherapy for breast cancer according to clinical guidelines. Treatment includes 8 cycles of chemotherapy administered every 3 weeks. No Traditional Chinese Medicine (TCM) is provided in this group.
  Groups: Conventional Western Medicine Treatment Group
Other: Integrative Treatment (Chemotherapy + TCM) — Participants in the integrative care group receive conventional chemotherapy combined with Traditional Chinese Medicine (TCM) treatment. Herbal formulas are prescribed by licensed TCM physicians based on syndrome differentiation and are aimed at strengthening vital qi and harmonizing stomach function. Treatment is conducted under Taiwan's National Health Insurance coverage.
  Groups: Integrative Treatment Group (Western Medicine + TCM)

SUMMARY:
The aim of this study is to investigate the intervention of traditional Chinese medicine (TCM) in managing the side effects experienced by breast cancer patients undergoing conventional Western medical treatments, such as blood cell decline, nausea, vomiting, gastrointestinal discomfort, and overall quality of life. The study aims to establish a long-term clinical enrollment criteria and process for TCM adjuvant therapy in breast cancer. The research design will utilize a prospective cohort study and real-world cross-sectional observational research method to obtain clinical data and survival status of the patients.

DETAILED DESCRIPTION:
Two-group parallel experimental design. One group received conventional Western medicine treatment, while the other group received combined treatment with both traditional Chinese and Western medicine treatment.

A. Patients who opt for integrated traditional Chinese medicine (TCM) treatment will be referred to the TCM outpatient department, where a TCM practitioner will prescribe TCM prescriptions, followed by the initial clinical effectiveness assessment.

B. Patients will continue their follow-up visits at the oncology and TCM clinics, receiving both conventional Western medicine treatments and TCM treatments.

C. Both the Western medicine treatments and TCM treatments received by the patients are covered by health insurance, and patients do not need to pay anyadditional fees.

D. Both the "Conventional Western Medicine Treatment Group" and the "Integrated Western and Chinese Medicine Treatment Group" will undergo another clinical effectiveness assessment (blood tests) before the next cancer treatment.

E. A questionnaire will be administered before starting chemotherapy and before each research visit for treatment evaluation. A final evaluation will be conducted within four weeks after the last radiation or chemotherapy session. The questionnaire includes the EOG, BFI-T, FACT-B,EORTC-QLQ-C30, EORTC-QLQ-BR23, WHOQOL-BREF, and BCQ.

ELIGIBILITY:
Inclusion Criteria:

* A. Aged 18 years or above.
* B. Female patients diagnosed with primary breast cancer and receiving Western medical treatment. The included breast cancer diagnosis codes based on ICD-9 are 174 to 179.

Exclusion Criteria:

* A. Patients with a prior diagnosis of other malignant tumors before being diagnosed with primary breast cancer.
* B. Patients with primary breast cancer who have not received Western medical treatment, meaning they have not undergone surgical resection, radiation therapy, chemotherapy, or targeted therapy..
* C. After taking Chinese medicine, those who have uncomfortable symptoms or whose behavior affects Western medicine treatment should withdraw from the trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — A. Aged 18 years or above.
  B. Female patients diagnosed with primary breast cancer and receiving Western medical treatment. The included breast cancer diagnosis codes based on ICD-9 are 174 to 179.
Study Population: Female breast cancer patients diagnosed by oncologists or surgeons at Taipei Tzu Chi Hospital, who are receiving or have received chemotherapy. Participants will be grouped based on their willingness to receive Traditional Chinese Medicine (TCM) in addition to standard Western medical treatment. All participants are aged 20 years or older and able to complete questionnaire-based assessments.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
FACT-B (Functional Assessment of Cancer Therapy - Breast) | A standard 8-cycle chemotherapy regimen will be administered every 21 days. Patient-reported outcome questionnaires will be collected at baseline (pre-Cycle 1), every other cycle , and 3 weeks after the final cycle.
  The FACT-B is a validated questionnaire used to assess quality of life in breast cancer patients. It includes domains such as physical well-being, social/family well-being, emotional well-being, functional well-being, and breast cancer-specific concerns.
EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30) | A standard 8-cycle chemotherapy regimen will be administered every 21 days. Patient-reported outcome questionnaires will be collected at baseline (pre-Cycle 1), every other cycle , and 3 weeks after the final cycle.
  The EORTC QLQ-C30 is a validated, cancer-specific, patient-reported quality of life questionnaire. It consists of 30 items covering five functional domains (physical, role, emotional, cognitive, and social), three symptom domains (fatigue, pain, nausea/vomiting), a global health status/QoL scale, and several single items (e.g., dyspnea, insomnia). It is widely used in cancer clinical trials for measuring changes in quality of life during treatment.
WHOQOL-BREF (World Health Organization Quality of Life - BREF) | A standard 8-cycle chemotherapy regimen will be administered every 21 days. Patient-reported outcome questionnaires will be collected at baseline (pre-Cycle 1), every other cycle , and 3 weeks after the final cycle.
  The WHOQOL-BREF is a 26-item questionnaire developed by the World Health Organization to assess an individual's perception of their quality of life in four domains: physical health, psychological health, social relationships, and environment. It is widely used for evaluating general quality of life in clinical populations.
BCQ (Body Constitution Questionnaire) | A standard 8-cycle chemotherapy regimen will be administered every 21 days. Patient-reported outcome questionnaires will be collected at baseline (pre-Cycle 1), every other cycle , and 3 weeks after the final cycle.
  The BCQ is a self-reported questionnaire developed based on Traditional Chinese Medicine (TCM) theory. It evaluates individual body constitution types, including Yang deficiency, Yin deficiency, and Stasis constitution. The tool is useful in assessing patients' constitutional status and monitoring changes during treatment, especially in integrative TCM studies.
EQ-5D (EuroQol Five Dimensions Questionnaire) | On the day of each chemotherapy cycle (Day 1 of each cycle)
  The EQ-5D is a standardized instrument developed by the EuroQol Group to measure health-related quality of life. It includes five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. It also includes a visual analog scale (VAS) to rate overall health. It is widely used in health economic evaluations and patient-reported outcome assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Hsien-Chang Wu, Principal Investigator — Taichung Tzu Chi Hospital
Locations (1):
- Buddhist Taipei Tzu Chi General Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data (IPD) will not be shared publicly. Data may be available upon reasonable request to the principal investigator after publication of the main study results, subject to approval of a data sharing agreement to protect participant privacy.